CLINICAL TRIAL: NCT03402542
Title: Eligibility Criteria for Cholecystectomy in Ambulatory Surgery
Status: Completed | Type: Observational
Sponsor: Pierre Wauthy (Other)
Responsible Party: Sponsor-Investigator, Pierre Wauthy, Head of clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-cholecystectomy
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Cholecystectomy
MeSH Terms: interventions — Cholecystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cholecystectomy: Patients with a symptomatic vesicular lithiasis, having undergone cholecystectomy during a scheduled hospitalization in the CHU Brugmann Hospital between May 2016 and November 2017.
  Interventions: Procedure: Cholecystectomy

INTERVENTIONS:
Procedure: Cholecystectomy — Cholecystectomy

SUMMARY:
Cold laparoscopic cholecystectomy is the gold standard for the management of symptomatic vesicular stones. There is considerable controversy as to whether it should be practiced in outpatient surgery or as part of inpatient surgery, regarding to patient safety.

"Minor" surgical procedures, such as anal surgery or simple inguinal hernia interventions, were initially considered eligible for an outpatient procedure. Advances in surgical techniques, anesthesia and early rehabilitation have also made it possible to consider more "heavy" interventions, such as cholecystectomy.

The aim of this study is to identify eligible patients for laparoscopic cholecystectomy in outpatient surgery, taking surgical criteria into account.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had a laparoscopic cholecystectomy with a single cholecystectomy procedure without other associated interventions (bariatric surgery or other)

Exclusion Criteria:

* Pregnant women
* Diabetic patients under insulin treatment
* History of major abdominal surgery
* Acute cholecystitis as per anatomo-pathological examination

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who have had a laparoscopic cholecystectomy with a single cholecystectomy procedure without other associated interventions (bariatric surgery or other). Hospitalisation within the CHU Brugmann Hospital between May 2016 and November 2017.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Surgery duration | Up to 4h
  Duration of the surgical intervention
Post surgical pain | Up to 1 day after surgery
  Pain killer medication administered post surgery, expressed in mg
Nausea | Up to 1 day after surgery
  Occurence of nausea or vomiting post surgery
Post surgery hospitalization duration | Up to 10 days after surgery
  Post surgery hospitalization duration
Medical complications after surgery | Up to 1 year after surgery
  Medical complications after surgery

SECONDARY OUTCOMES:
Data extraction from medical files: medical history | 5 min
  Important surgical or medical antecedents of the patient before surgery (data extraction from medical file).
Physical status score | 5 min
  Physical status score (also called ASA score for American Society of Anesthesiologists score) of the patient before surgery. The ASA score ranges from I (normal healthy patient) to VI (declared brain-dead patient whose organs are being removed for donor purposes)
Body mass index | 5 min
  Body mass index of the patient before surgery
Hospitalisation type | Up to 10 days after surgery
  Same day (ambulatory) or not
Type of surgery | Up to 4 hours
  Surgery performed under nuclear magnetic resonance (RMN) or RMN + endoscopic retrograde cholangiography (CWR)

CONTACTS AND LOCATIONS:
Overall Officials: Levon HAKOBYAN, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No